CLINICAL TRIAL: NCT00447837
Title: A Phase 2, Double-Blind, Placebo-Controlled, Multi-Center, Randomized Study Evaluating the Safety and Efficacy of SPRC-AB01, Tobramycin Solution for Nasal Inhalation, in Post-Surgical Subjects With Chronic Sinusitis
Brief Title: Evaluating SPRC-AB01 in Post-Surgical Subjects With Chronic Sinusitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Naryx Pharma (Industry)
Responsible Party: Kimberly Salgado/VP Product Development, Naryx Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPRC-AB01-003
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2007-12

CONDITIONS: Chronic Sinusitis
Keywords: Chronic Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: SPRC-AB01
- 2 (Experimental)
  Interventions: Drug: SPRC-AB01
- 3 (Placebo Comparator)
  Interventions: Drug: SPRC-AB01

INTERVENTIONS:
Drug: SPRC-AB01 — 90 mg/3 mL BID, 180 mg/3 mL bid, placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and efficacy of SPRC-AB01 versus placebo for treatment of chronic sinusitis in subjects who have had sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient subjects who have signed a written informed consent.
* A documented history of chronic sinusitis with clinical signs and symptoms suggestive of inflammation or infection for at least 90 consecutive days.
* A documented history of sinus surgery > 90 days.
* Nasal endoscopic exam documenting purulence (pus) from an open sinus cavity with mucosal swelling/edema.
* Women of childbearing potential must have a negative serum pregnancy test and must use adequate birth control throughout the study.

Exclusion Criteria:

* Pregnant females and females unwilling to use adequate birth control.
* Use of any investigational drug/device within 30 days of study screening.
* The following medications will require a certain washout period as determined by the protocol: systemic corticosteroids, mast cells and/or leukotriene inhibitors, anti-inflammatories, decongestants, antihistamines, non-steroidal anti-inflammatory (NSAID) or cyclooxygenase (COX)-2 inhibitors, antibiotics or antifungals.
* Presence of other infections which may require use of systemic antibiotics.
* Known allergy or hypersensitivity to aminoglycosides or other study drug formulation components.
* Recent hospitalization for any reason and/or major surgeries within 30 days of study screening.
* Major elective and/or nasal and/or sinus surgical procedures (including sinuplasty) within 90 days before or 90 days after study screening.
* Known history of neurological or muscular disorders.
* Diagnosis of an immunodeficiency disease.
* Previous diagnosis of cystic fibrosis, ciliary dyskinesias, Kartagener syndrome, empty nose syndrome, Wegener granulomatosis, Churg-Strauss syndrome, Samter syndrome, or sarcoidosis.
* Current or known history of tinnitus, vertigo, or significant sensorineural hearing loss.
* Recent history of alcohol or drug abuse.
* Inability to understand the nature, scope, and possible consequences of the study or study procedures, unless cared for by a legally authorized representative.
* Inability to adhere to the study requirements.
* Previous participation in any Naryx Pharma protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in TSSS during first week post-therapy | 86 days

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Clinical Research Consultants, Hoover, Alabama
  - NEA Clinic, Jonesboro, Arkansas
  - Central California Clinical Research, Fresno, California
  - Allergy Research Foundation, Inc, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Allergy Medical Group of the North Area Inc, Roseville, California
  - Sacramento Ear, Nose & Throat, Sacramento, California
  - Allergy & Asthma Medical Group and Research Center, San Diego, California
  - 1st Allergy & Clinical Research Center, Centennial, Colorado
  - Colorado Otolaryngology Associates, Colorado Springs, Colorado
  - The Connecticut Sinus Center, Bridgeport, Connecticut
  - Clinical Trials Management LLC, Boca Raton, Florida
  - Allergy & Asthma Center / South Florida ENT, Fort Lauderdale, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Nasal Sinus and Allergy Institute, Alpharetta, Georgia
  - Northeast Georgia Research Center, Gainsville, Georgia
  - Northside Ear, Nose & Throat, Roswell, Georgia
  - Commonwealth Ear, Nose & Throat, Louisville, Kentucky
  - Calvert Internal Medicine Group, Prince Frederick, Maryland
  - Massachusetts General Hospital - Allergy Clinical Research, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Clinical Research Institute, Plymouth, Minnesota
  - Allergy & Sinus Center, Greenwood, Mississippi
  - Clinical Research Group of Montana, Bozeman, Montana
  - Shah Eye Ear Nose & Throat, Lawrenceville, New Jersey
  - ENT Care, Somerville, New Jersey
  - Weill Medical College-Department of Otorhinolaryngology, New York, New York
  - University of Rochester-Otolaryngology Associates, Rochester, New York
  - Center for Allergy and Asthma of Bronx and Westchester, The Bronx, New York
  - Charlotte Eye, Ear, Nose & Throat Associates, Charlotte, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Cleveland Clinic - Head & Neck Institute, Cleveland, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - University of Pittsburgh - The Eye and Ear Institute, Pittsburgh, Pennsylvania
  - ADAC Research PA, Greenville, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - The Allergy, Asthma & Sinus Center, Knoxville, Tennessee
  - Ear, Nose & Throat Associates of Corpus Christi / Research, Corpus Christi, Texas
  - Allergy and Asthma Associates, Houston, Texas
  - Research Across America, Plano, Texas
  - San Antonio Ear, Nose and Throat Research, San Antonio, Texas
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin